CLINICAL TRIAL: NCT07028879
Title: Effectiveness of a One-year Group Program for Fatigue Management in Minimally Impaired People With Multiple Sclerosis: a Non-randomized, Open-label, Controlled Clinical Trial
Brief Title: Effectiveness of a One-year Group Program for Fatigue Management in Minimally Impaired People With Multiple Sclerosis
Acronym: HCB_MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HCB/2025/0049
Record Dates: First submitted 2025-05-23; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Combination of Occupational Therapy and Physiotherapy strategies and sessions in-person, 2 days-week, during 12 months.
  Interventions: Procedure: Fatigue management program
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Fatigue management program — Combination of Occupational Therapy and Physiotherapy strategies and sessions.
  Arms: Intervention group

SUMMARY:
Fatigue is one of the most common symptoms, experienced by between 50% and 100% of people with multiple sclerosis (MS), and contributes significantly to the consequences of MS and perceived disability in the daily lives of those with the condition. On the one hand, practicing different forms of physical exercise (PE) has demonstrated effective management of perceived fatigue, and the literature strongly supports the need for regular exercise in patients with MS.

On the other hand, energy conservation programs and cognitive-behavioral interventions have demonstrated improvements in self-efficacy, participation in social life, perceived control over their disease, and a reduction in the perceived impact of fatigue, particularly in the physical and psychosocial domains of life.

Therefore, in this study, a physical therapist and an occupational therapist will conduct a one-year group program focused on educational and practical learning of techniques and strategies, keeping in mind that lifestyle changes take time to become permanent.

It is important to highlight that, as MS generally presents in early adulthood, there is growing interest in exploring rehabilitation techniques very early after diagnosis or in minimally affected MS patients (0-4.5 on the EDSS), we are therefore interested in exploring this program in this population group with MS, the majority of whom are actively employed, and evaluating the effects on perceived fatigue severity, quality of life, incidental and planned exercise, sleep quality, anxiety and depression, and perceived self-efficacy.

Study participants will be recruited by the neuroimmunology team at Hospital Clínic de Barcelona, who will select those who meet the inclusion criteria from the multiple sclerosis patients seen. Those patients who, despite meeting the inclusion criteria, are unable to attend the sessions (due to availability, geographic location, or other personal reasons) will form the comparison group. Therefore, there is no random assignment in this study. For this study, a total sample of 28 patients will be divided into three groups of 7, 7, and 14 participants, respectively. The last group will not receive treatment and will be used as a control group. Patients who do receive treatment will be assigned to groups on a first-come, first-served basis, and the therapeutic program will be the same for both groups. This separation is done to improve the quality of the intervention by allowing participants greater interaction in small groups.

Participants who must withdraw from the study for reasons beyond their control, having completed less than a third of the program, and participants who, despite being considered good candidates, are unable to attend the sessions for work, personal, or geographic reasons, will be evaluated at the beginning and end of the study using the same scales as the control group to compare the results obtained.

The sessions will be held at the day hospital for neurodegenerative diseases at the Hospital Clínic de Barcelona, twice a week: one physiotherapy session and one occupational therapy session. Implicit assessments will be conducted at the start of the program, at 6 months, one year, and 6 months after completion of the program.

There are no risks beyond the risks inherent in sports practice, which may exist in physical therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple sclerosis referred by the Neuroimmunology and Multiple Sclerosis Unit at Hospital Clínic de Barcelona who present symptoms of limiting fatigue.
* Independence to perform basic activities of daily living.
* Maximum EDSS score of 4.5.

Inclusion criteria for control group participants:

* Patients who, despite meeting the inclusion criteria (6.1), are unable to attend the sessions (due to availability, geographic location, or other personal reasons) will be included in the comparison group. or
* Those who show a lack of attendance at sessions of <80% over the course of a year or <75% in one of the quarters.

Exclusion Criteria:

* Severe comorbidity due to other conditions, including severe depressive symptoms, or substance use that may impact the individual's self-perception.
* MS flare within 30 days prior to inclusion.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-09-13 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in reducing the severity of perceived fatigue by the Modified Fatigue Impact Scale (MFIS). | (12 months after the start of the program) and at mid-term follow-up (18 months)
  This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items. The abbreviated version can be used if time is limited, but the full-length version has the advantage of generating subscales. Administration time is approximately 5-10 minutes for the full-length version and 2-3 minutes for the abbreviated version. The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument. The total score for the MFIS is the sum of the scores for the 21 items.

SECONDARY OUTCOMES:
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in improving self-efficacy by the 4-item Spanish chronic disease self - efficacy. | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The four-item Spanish-language version (SEMCD-S) was developed to measure changes in self-efficacy in program participants and have been used in a numerous evaluations of chronic disease self-management programs. The score for each item is the number circled. If two consecutive numbers are circled, code the lower number (less self-efficacy). If the numbers are not consecutive, do not score the item. The score for the scale is the mean of the eight items. If more than two items are missing, do not score the scale. Higher number indicates higher self-efficacy.
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in improving incidental and planned exercise by the International Physical Activity Questionnaire (IPAQ) | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The International Physical Activity Questionnaire (IPAQ) measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. Test score:
  1. Vigorous physical activity: 8 METs x minutes x days per week
  2. Moderate physical activity: 4 METs x minutes x days per week
  3. Walking: 3.3 x minutes x days per week.
  Then add the three values obtained:
  TOTAL = Vigorous physical activity + Moderate physical activity + walking
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in improving sleep quality by the Pittsburgh Sleep Quality Index (PSQI). | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Scoring the PSQI: each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in Reducing anxiety and depression levels by the Hospital Anxiety and Depression Scale (HADS). | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale, with seven items relating to anxiety and seven relating to depression. It was created to measure specifically to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness, for example fatigue and insomnia or hypersomnia. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in reducing the impact of fatigue on health status by the EQ-5D-5L. | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The EQ-5D-5L is a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state; EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
To determine the effectiveness of this program after completion (12 months after the start of the program) and at mid-term follow-up (18 months) in improving quality of life by the SF-36 questionnaire. | (12 months after the start of the program) and at mid-term follow-up (18 months)
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life. It measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: No